CLINICAL TRIAL: NCT03728829
Title: An Observational Phase II Trial of Targeted Next Generation Sequencing Analysis for the Efficacy of Trastuzumab Neoadjuvant Chemotherapy in Patients With HER2 Positive Breast Cancer
Brief Title: Targeted Next Generation Sequencing for the Efficacy of Trastuzumab Neoadjuvant Chemotherapy in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: OrigiMed (Industry)
Responsible Party: Principal Investigator, Liu Yunjiang, Vice President, Clinical Professor, Hebei Medical University Fourth Hospital
Other Study IDs: YLiu
Record Dates: First submitted 2018-10-26; First posted 2018-11-02 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Observational; Prospective
Keywords: breast cancer; HER2 positive; next generation sequencing; trastuzumab; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained, with potential for extraction of DNA from at least one of the types of samples retained (tissue, whole blood)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trastuzumab+TP neoadjuvant chemotherapy: 100 cases of patients with stage II-III HER2+ breast cancer will be assigned participants to neoadjuvant treatment regimen, including Trastuzumab combined with Docetaxel and Carboplatin. 5-10 ml peripheral blood will be collected from each patient and formalin fixed paraffin embedded (FFPE) blocks/sections or fresh tumor tissues/biopsies will be obtained from the hospitals before and after neoadjuvant therapy. The genomic characteristics between patients achieved pCR and non-pCR will be analyzed. The clinically actionable mutations for future therapy instructions will be identified.
  Interventions: Drug: Trastuzumab+TP

INTERVENTIONS:
Drug: Trastuzumab+TP — Trastuzumab (4 mg/kg loading dose, then 2 mg/kg I.V., every week, totally 17 weeks (6 cycles)) combined with TC neoadjuvant chemotherapy (Docetaxel 75 mg/m2 I.V., day 1, Carboplatin 400 mg/kg, I.V., day 2, every 3 weeks, totally 6 cycles).
  Other Names: Trastuzumab+Docetaxel+Carboplatin

SUMMARY:
To explore the genetic background of patients with HER2 positive breast cancer that benefit from trastuzumab combined with neoadjuvant chemotherapy, identify clinically actionable mutations that associated with trastuzumab resistance or drug efficacy, we designed this Observational phase II trial. The primary endpoint is genetic profile of HER2+ breast cancer patients treated with trastuzumab combined neoadjuvant chemotherapy. Secondary endpoints included pathological complete response (pCR) rate and safety.

DETAILED DESCRIPTION:
Currently, patients with stage II-III breast cancer still accounts for a large population in China, and neoadjuvant therapy is considered the standard treatment for them. The pathological complete response (pCR) rate takes for an indicator for regimens efficacy, and the achievement of pCR after neoadjuvant chemotherapy is associated with favorable outcomes including disease-free survival and overall survival.

HER2+ breast cancer represents an invasive and poor prognosis subtype, and the efficacy of neoadjuvant therapy for these patients has been greatly augmented by the addition of trastuzumab. However, more than 50% of HER2+ breast cancer patients treated with trastuzumab combined neoadjuvant chemotherapy cannot achieve pCR, even experience primary drug resistance and rapid disease progression. Therefore, to explore the genomic features of the population that benefited from trastuzumab combined with chemotherapy is of great significance for personalized treatment of HER2+ breast cancer, aiming to avoid overtreatment and identify clinically actionable mutations for future therapy instructions.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-70 years old at the time of diagnosis of primary breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1
* Stage III breast cancer according to the 7th Edition of Cancer staging Manual of American Joint Committee on Cancer (AJCC)
* full assessment of ER, PR and HER2 status of primary tumor in accordance with the American Society of Clinical Oncology (ASCO) guidelines
* pathological diagnosis and all courses of treatment confirmed

Exclusion Criteria:

* any known metastatic disease, by physical exam or by imaging studies such as computed tomography (CT)/magnetic resonance imaging (MRI), at the time of study entry
* any previous exposure to chemotherapy, radiotherapy, or endocrine therapy
* left ventricular ejection fraction (LVEF) < 55% by Echocardiogram (ECHO) or multigated acquisition scan (MUGA) or significant clinical symptoms or signs of heart failure
* major organ dysfunction, inclusive of bone marrow, renal, liver and hepatic function, that would prohibit patients from receiving standard chemotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
genetic profile sequenced by a pan-cancer gene panel | 1 year
  analyze the genetic profile of HER2+ breast cancer patients treated with trastuzumab combined neoadjuvant chemotherapy by targeted next generation sequencing on a pan-cancer gene panel

SECONDARY OUTCOMES:
pCR | 1 year
  The pathological complete response (pCR) rate of patients treated with trastuzumab neoadjuvant chemotherapy.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 year
  The incidence of adverse events of patients treated with trastuzumab neoadjuvant chemotherapy, including Cardiac toxicity, leukopenia, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Baoen Shan, MD,PhD, Study Chair — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, China, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No